CLINICAL TRIAL: NCT02811796
Title: Prospective Validation of the Angio-based Fractional Flow Reserve (Quantitative Flow Ratio, QFR) System to Discriminate Patients at Risk of Adverse Events After Stent Implantation.
Brief Title: Angio-based Fractional Flow Reserve to Predict Adverse Events After Stent Implantation
Acronym: HAWKEYE
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, Interventional Cardiologist, University Hospital of Ferrara
Other Study IDs: 190678
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Prognosis; Stents
Keywords: drug eluting stents; flow fractional reserve; prognosis; angio-based FFR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- angio-based FFR estimation: The investigators will include all patients receiving successful coronary stent implantation. In these patients the investigators will acquire specific angiograms to permit angio-based FFR (QFR) calculation. An independent corelab will estimate the QFR value. This value will be related to prognosis to verify if it is able to discriminate those at higher risk of adverse events.
  Interventions: Other: angio-based FFR estimation

INTERVENTIONS:
Other: angio-based FFR estimation — The investigators will acquire specific angiograms to permit angio-based FFR (QFR) calculation. An independent corelab will estimate the QFR value. This value will be related to prognosis to verify if it is able to discriminate those at higher risk of adverse events.

SUMMARY:
The investigators will collect prospectively baseline, procedural and follow-up data of all patients receiving successful percutaneous coronary intervention (PCI) and stent implantation. Angio-based flow fractional reserve (quantitative flow ratio, QFR, Medis medical imaging systems Leiden, The Netherlands) will be estimated in all patients. Especially, the investigators at the end of the procedure (this is defined according operator's judgement) will record 2 orthogonal angiograms (as suggested by QFR instructions) at 15 frames/second and the same 2 orthogonal angiograms at 30 frames/second. An independent corelab (blinded to procedural data and clinical outcome) will estimate QFR value (one with the angiograms at 15 frames and one with those at 30 frames

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) allows to evaluate the functional significance of coronary artery lesions, through the ratio of the mean coronary artery pressure after the stenosis to the mean aortic pressure during maximum hyperaemia. The actual widely accepted cutoff value is 0.80. Below this value, an intermediate coronary lesion is considered significant and its treatment with percutaneous coronary intervention (PCI) is justified.

The measurement FFR after stent implantation has a strong predictive value with respect to death, myocardial infarction, or need for repeat revascularization of the target vessel within 6 months. The higher the FFR, the lower the event rate. FFR cut-off of 0.90 might be a useful indicator in daily practice for optimal physiologic stent implantation. Nevertheless, the use of the FFR in the post stenting , is relatively low, because of costs of the pressure wire and the adverse effects related to the use of adenosine.

A new method (QFR by Medis medical imaging) for evaluation of the functional significance of coronary stenosis is based on computer calculation of the FFR value. This calculation is performed by analysing the coronary angiogram and thus reduces or potentially eliminates the need for measuring FFR by pressure wires. The QFR method combines a 3D reconstructions of the target vessel based on two angiographic projections and the contrast flow velocity to compute the "FFR value". To perform QFR the investigators will acquire two angiographic projections with angle >25 degree that allow the 3D reconstruction of the vessel (see values below).

Projections for left main (LM) and proximal left anterior descending (LAD) or proximal left circumflex (LCX): right anterior oblique (RAO) 20, Caudal 45 and anterior-posterior (AP), Caudal 10

Projections for LAD/diagonal: AP, Cranial 45 and RAO 35, Cranial 20

Projections for LCX/obtuse marginal (OM): left anterior oblique (LAO) 10, Caudal 45 and RAO 25, Caudal 25

Projections for Proximal+Mid right coronary artery (RCA): LAO 45, caudal (CAUD) 0 and AP, CAUD 0

Projections for postero-lateral artery and posterior-descending artery (PLA/PDA): LAO 45, CAUD 0 and LAO 30, CAUD 30

Finally, the investigators will assess the relationship between QFR value and adverse events. We will assess the best QFR value able to discriminate the cumulative occurrence of adverse events. In the study, we will include also ST-segment elevation myocardial infarction patients. This subset of patients will be analysed as independent cohort to obtain preliminary results and will be analysed in a independent study

ELIGIBILITY:
Inclusion Criteria:

-successfull percutaneous coronary intervention and stent implantation

Exclusion Criteria:

* inability to provide consent
* inability to guarantee at least 1-year follow-up
* thrombolysis in myocardial infarction (TIMI) flow <3
* life expectancy <1 year
* previous coronary artery bypass graft
* atrial fibrillation
* ongoing ventricular arrhythmias
* significant and persistent tachycardia (heart rate >100 bpm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receiving complete revascularization with successful PCI and stent implantation (second generation drug eluting stent)
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Device-oriented cardiac events | 1-year
  cumulative occurrence of cardiac death, target vessel myocardial infarction, target lesion revascularization

SECONDARY OUTCOMES:
cardiac death | 1-year
  cumulative occurrence of cardiac death
all-cause mortality | 1-year
  cumulative occurrence of all-cause mortality
any myocardial infarction | 1-year
  cumulative occurrence of any myocardial infarction
target vessel revascularization | 1-year
  cumulative occurrence of target vessel revascularization
stent thrombosis | 1-year
  cumulative occurrence of definite, probable and possible stent thrombosis
hospital admission for all causes | 1-year
  cumulative occurrence of hospital admission for all causes

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (6):
  - University Hospital of Ferrara, Cona, Ferrara
  - ASP Agrigento, Agrigento
  - Ospedale Civile, Agrigento
  - Caserta
  - San Luigi Gonzaga, Orbassano
  - Ospedale Civile, Seriate
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Biscaglia S, Uretsky BF, Tebaldi M, Erriquez A, Brugaletta S, Cerrato E, Quadri G, Spitaleri G, Colaiori I, Di Girolamo D, Scoccia A, Zucchetti O, D'Aniello E, Manfrini M, Pavasini R, Barbato E, Campo G. Angio-Based Fractional Flow Reserve, Functional Pattern of Coronary Artery Disease, and Prediction of Percutaneous Coronary Intervention Result: a Proof-of-Concept Study. Cardiovasc Drugs Ther. 2022 Aug;36(4):645-653. doi: 10.1007/s10557-021-07162-6. Epub 2021 Apr 8. PMID 33830399
- [Derived] Biscaglia S, Tebaldi M, Brugaletta S, Cerrato E, Erriquez A, Passarini G, Ielasi A, Spitaleri G, Di Girolamo D, Mezzapelle G, Geraci S, Manfrini M, Pavasini R, Barbato E, Campo G. Prognostic Value of QFR Measured Immediately After Successful Stent Implantation: The International Multicenter Prospective HAWKEYE Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2079-2088. doi: 10.1016/j.jcin.2019.06.003. Epub 2019 Sep 25. PMID 31563688